CLINICAL TRIAL: NCT05047263
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Phase 3 Study to Investigate the Efficacy and Safety of FInerenone, in Addition to Standard of Care, on the Progression of Kidney Disease in Patients With Non-Diabetic Chronic Kidney Disease
Brief Title: A Trial to Learn How Well Finerenone Works and How Safe it is in Adult Participants With Non-diabetic Chronic Kidney Disease
Acronym: FIND-CKD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21177; 2021-000421-27 (EudraCT Number)
Record Dates: First submitted 2021-09-12; First posted 2021-09-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non-diabetic Chronic Kidney Disease
MeSH Terms: interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Finerenone (BAY94-8862) (Experimental): Participants will receive finerenone.
  Interventions: Drug: Finerenone (BAY94-8862)
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone (BAY94-8862) — Tablet, 10 mg or 20 mg, once daily (OD), oral
  Arms: Finerenone (BAY94-8862)
Drug: Placebo — Tablet, once daily, oral
  Arms: Placebo

SUMMARY:
Researchers are looking for a better way to treat people who have non-diabetic chronic kidney disease (non-diabetic CKD). The trial treatment, finerenone, is being developed to help people who have long lasting kidney disease, also known as chronic kidney disease (CKD). It works by blocking a certain hormone called aldosterone that causes injury and inflammation in the heart and kidney which is known to play a role in CKD.

In this trial, the researchers want to learn if finerenone helps to slow down the worsening of the participants' non-diabetic CKD compared to a placebo. A placebo looks like a trial treatment but does not have any medicine in it. The trial will include about 1,580 men and women who are at least 18 years old.

The participants will take finerenone or a placebo once a day as tablets by mouth. All of the participants will also continue to take their current medicine for their CKD. The participants will be in the trial for up to about 50 months.

During the trial, the doctors will collect blood and urine samples and check the participants' health. The participants will also answer questions about how they are feeling and what adverse events they are having. An adverse event is a medical problem that happens during the trial. Doctors keep track of all adverse events that happen in trials, even if they do not think the adverse events might be related to the trial treatments.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of chronic kidney disease and:

  * Urine albumin/creatinine ratio (UACR) of ≥ 200 but ≤ 3500 mg/g and estimated glomerular filtration rate (eGFR) ≥ 25 but < 90 mL/min/1.73m^2 at screening, and
  * Documentation of albuminuria/proteinuria in the participant's medical records at least 3 months prior to screening.
* Stable and maximum tolerated labeled dose of an Angiotensin-converting enzyme inhibitor (ACEI) or Angiotensin receptor blocker (ARB) for at least 4 weeks prior to screening
* K+ ≤ 4.8 mmol/L at screening

Exclusion Criteria:

* Established diagnosis of Type 1 or 2 Diabetes mellitus, or HbA1c ≥ 6.5% (48 mmol/mol)
* Autosomal dominant or autosomal recessive polycystic kidney disease
* Lupus nephritis or anti-neutrophilic cytoplasmic autoantibody (ANCA) -associated vasculitis or any other primary or secondary kidney disease requiring immunosuppressive therapy within 6 months prior to screening
* Symptomatic heart failure with reduced ejection fraction with class 1A indication for Mineralocorticoid receptor antagonists (MRAs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1584 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
Mean rate of change as measured by the total slope of eGFR from baseline to Month-32. | From baseline to month 32
  eGFR: Estimated glomerular filtration rate

SECONDARY OUTCOMES:
Time to the composite of kidney failure, sustained eGFR decline of >= 57%, heart failure hospitalization or Cardiovascular (CV) death | Up to end of study visit (up to approximately 49 months)
Time to the composite of kidney failure or sustained eGFR decline of >= 57% | Up to end of study visit (up to approximately 49 months)
Time to the composite to heart failure hospitalization or CV death | Up to end of study visit (up to approximately 49 months)
Number of participants with Treatment-emergent adverse events (TEAEs), Treatment-emergent serious adverse events (TESAEs) and Adverse events of special interest (AESI) | Up to approximately 50 months

CONTACTS AND LOCATIONS:
Locations (326):
- United States (57):
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - Balboa Research SMO+ - Chula Vista - West, Chula Vista, California
  - Balboa Research SMO+ - El Centro, El Centro, California
  - UCLA Clinical and Translational Research Center - Nephrology, Los Angeles, California
  - Balboa Nephrology Medical Group - Poway, Poway, California
  - North America Research Institute - San Dimas, San Dimas, California
  - United Clinical Research & Innovations, South Gate, California
  - University of Colorado | Renal Research Office, Aurora, Colorado
  - DaVita Clinical Research | Middlebury, CT, Middlebury, Connecticut
  - Yale University | Nephrology Clinical Research, New Haven, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Research Physicians Network Alliance, Boca Raton, Florida
  - Florida Kidney Physicians - Boca Raton, Boca Raton, Florida
  - AdventHealth Translational Research Institute, Orlando, Florida
  - Grady Memorial Hospital - Endocrinology, Atlanta, Georgia
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - Central Georgia Kidney Specialists - Macon, Macon, Georgia
  - Frenova Renal Research | Boise Kidney and Hypertension, Meridian, Idaho
  - Northwestern Medicine - Feinberg School of Medicine - Nephrology and Hypertension, Chicago, Illinois
  - Research by Design, LLC | Chicago, IL, Chicago, Illinois
  - Nephrology Associates of Northern Illinois and Indiana - Hinsdale, Hinsdale, Illinois
  - University of Iowa Health Care Medical Center - Cardiology, Iowa City, Iowa
  - KUMC Clinical and Translational Science Unit - Nephrology, Kansas City, Kansas
  - Kansas Nephrology Research Institute, Wichita, Kansas
  - Wichita Nephrology Group, PA, Wichita, Kansas
  - Northwest Louisiana Nephrology - Shreveport - 1800 Buckner St., Shreveport, Louisiana
  - Johns Hopkins Hospital - Nephrology, Baltimore, Maryland
  - Tufts Medical Center | Nephrology Department, Boston, Massachusetts
  - DaVita Clinical Research | Edina, MN, Edina, Minnesota
  - University Hospital - UMMC - Nephrology, Jackson, Mississippi
  - Clinical Research Consultants, a JCCT Company, Kansas City, Missouri
  - St. Louis Heart and Vascular, PC - Christian Hospital Office, St Louis, Missouri
  - UNM Clinical and Translational Science Center - Nephrology, Albuquerque, New Mexico
  - Mountain Kidney & Hypertension Associates, Asheville, North Carolina
  - UNC Hospitals Outpatient Center at Eastowne - Nephrology, Chapel Hill, North Carolina
  - East Carolina University | Nephrology & Hypertension, Greenville, North Carolina
  - Eastern Nephrology Associates | Wilmington, Wilmington, North Carolina
  - UH Cleveland Medical Center - Nephrology, Cleveland, Ohio
  - Cleveland Clinic | Urological and Kidney Department, Cleveland, Ohio
  - Northeast Clinical Research Center | Bethlehem, PA, Bethlehem, Pennsylvania
  - Geisinger Medical Center - Nephrology, Danville, Pennsylvania
  - Temple Health - Nephrology, Philadelphia, Pennsylvania
  - South Carolina Clinical Reserach, Orangeburg, South Carolina
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Vanderbilt University Medical Center - Nephrology Clinical Trials Center, Nashville, Tennessee
  - Dallas Renal Group - Medical City, Dallas, Texas
  - El Paso Medical Research Institute (MedResearch Inc) | El Paso, TX, El Paso, Texas
  - DaVita Clinical Research | Houston, TX, Houston, Texas
  - Gamma Medical Research, Inc., McAllen, Texas
  - Texas Diabetes Institute - Renal Clinic, San Antonio, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - DaVita Clinical Research | North Houston, TX, Shenandoah, Texas
  - University of Utah School of Medicine | Kidney Research Clinic, Salt Lake City, Utah
  - Utah Kidney Research Institute | Salt Lake City, UT, South Salt Lake, Utah
  - Nephrology Associates of Northern Virginia - Fair Oaks, Fairfax, Virginia
  - Mendez Center For Clinical Research | Woodbridge, VA, Woodbridge, Virginia
  - Providence Medical Research Center, Spokane Valley, Washington
- Argentina (10):
  - Asociacion de Fomento y Sala de Primeros Auxilios Alberto Mignaburu | Berazategui, Argentina, Berazategui, Buenos Aires
  - Centro de Investigaciones Metabolicas | Ciudad de Autonoma de Buenos Aires, Argentina, Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Centro de Investigaciones Medicas Lanus | Buenos Aires, Argentina, Lanús, Buenos Aires
  - Instituto de Investigaciones Clinicas de Mar del Plata | Mar del Plata, Argentina, Mar del Plata, Buenos Aires
  - CEDIC Centro de Investigación Clínica | Buenos Aires, Argentina, CABA, Ciudad Auton. de Buenos Aires
  - Centro de Rehabilitacion Cardiovascular | San Luis, Argentina, San Luis, San Luis Province
  - Centro de Investigación y Prevención Cardiovascular, Buenos Aires
  - Clinica Privada Velez Sarsfield, Córdoba
  - Clinica de Nefrologia Urologia y Enfermedades Cardiovascular, Santa Fe
  - Centro de Investigaciones Clinicas del Litoral | Santa Fe, Argentina, Santa Fe
- Australia (8):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Illawarra Shoalhaven Local Health District, Wollongong, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Princess Alexandra Hospital Australia, Woolloongabba, Queensland
  - Eastern Health Integrated Renal Service, Box Hill, Victoria
  - Melbourne Renal Research Group, Reservoir, Victoria
  - Sunshine Hospital, St Albans, Victoria
- Belgium (6):
  - AZ Groeninge Campus Kennedylaan | Nephrology, Kortrijk, West-Vlaanderen
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liège, Liège
  - AZ Delta / Nephrology, Roeselare
- Bulgaria (8):
  - Medical Center ''4Life'', Burgas
  - Viva Phoenix Medical Center | Clinical Trials Department, Dobrich
  - Multiprofile Hospital for Active Treatment St. Ivan Rilski - Gorna Oryahovitsa | Nephrology Department, Gorna Oryahovitsa
  - Medical Center Hera | Montana Branch, Montana
  - Multiprofile Hospital for Active Treatment Sveti Georgi OOD, Pernik - Department of Cardiology, Pernik
  - Diagnostic-Consultative Center XX | Nephrology Department, Sofia
  - Medical Center Zara-Med EOOD | Nephrology Department, Stara Zagora
  - Medical Center ''Nevromedics'', Veliko Tarnovo
- China (45):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Second Hospital of Anhui medical university, Hefei, Anhui
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of TCM, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Jiangmen Wuyi Hospital of traditional Chinese Medicine, Jiangmen, Guangdong
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - People's Hospital of Liuzhou City, Liuchow, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The First affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Wuhan Hospital Of Traditional Chinese And Western Medicine, Wuhan, Hubei
  - Puai Hospital,Tongji Medical College, Huazhong Univ Sci&Tech, Wuhan, Hubei
  - Renmin Hosp., Wuhan Univ., Wuhan, Hubei
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - 1st Peopl's Hosp of Changzhou 3rd Affil Hosp of Soochow Univ, Changzhou, Jiangsu
  - Huai'an First People's Hospital, Nanjing Medical University, Huai'an, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - Jiangxi PingXiang people's Hospital, Pingxiang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Siping Central Hospital, Siping, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qilu Hosp., Shandong Univ., Jinan, Shandong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - SichuanAcademyofMedicalSciences&SichuanProvincialPeople'sHos, Chengdu, Sichuan
  - Sichuan University West China Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Hwa Mei Hospital, University of Chinese Academy Sciences, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical Univ (New), Wenzhou, Zhejiang
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Daping Hospital, 3rd Affil Hosp. 3rd Military Med Univ PLA, Chongqing
  - Zhongshan Hospital, Fudan University - Oncology Department, Shanghai
  - Xinhua Hos Affiliated to SH Jiaotong Uni School of Medicine, Shanghai
  - Shanghai Fifth People's Hospital,Fudan University, Shanghai
  - Central Hospital of Minhang District, Shanghai, Shanghai
  - Tianjin Union Medicine Centre (People's Hospital of Tianjin), Tianjin
- Czechia (10):
  - Fakultní nemocnice Brno - Interní gastroenterologická klinika, Brno, South Moravian
  - MUDr.Petr Bucek s.r.o., Frýdek-Místek
  - CTC Hodonín, s.r.o., Hodonín
  - Fakultni nemocnice Ostrava, Ostrava
  - Privamed s.r.o., Pilsen
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Nefrologicka ambulance, Prague
  - Nefromed s.r.o., Prague
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
  - Nemocnice Znojmo, Znojmo
- Denmark (6):
  - Rigshospitalet, Copenhagen University Hospital | Department of Nefrology, Copenhagen
  - Hospital of South West Jutland | Department of Endocrinology Research, Esbjerg
  - Herlev Hospital | Nephrology Department, Herlev
  - Region Midtjylland | Regionshospitalet Godstrup - Nephrology Department, Herning
  - Region Sjælland | Holbaek Sygehus - Cardiology department, Holbæk
  - Odense University Hospital | Department of Kidney Medicine, Odense C
- Greece (9):
  - General Hospital of Arta | Nephrology Department, Arta
  - HIPPOKRATION General Hospital of Athens, Athens
  - General Hospital of Athens LAIKO, Athens
  - General Hospital Of Thessaloniki Papageorgiou-Renal Department, Efkarpia
  - University General Hospital of Heraklion-Nephrology Clinic, Heraklion
  - University General Hospital Of Ioannina-Nephrology Clinic, Ioannina
  - University General Hospital of Patras | Nephrology Clinic, Pátrai
  - Ippokratio General Hospital Of Thessaloniki- 1st Department of Nephrology, Thessaloniki
  - Geniko Nosokomeio Thessalonikis George Papanikolaou-Nephrology Department, Thessaloniki
- Hong Kong (4):
  - Tung Wah Hospital, Sheung Wan, Hong Kong Island
  - Prince of Wales Hospital, Hong Kong, Hong Kong SAR
  - Princess Margaret Hospital, Hong Kong, Hong Kong SAR
  - Queen Mary Hospital, Hong Kong, Hong Kong SAR
- Hungary (7):
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai és Infektologiai Intezet, Budapest
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa
  - Nagykanizsai Kanizsai Dorottya Korhaz, Nagykanizsa
  - Medifarma-98 Egeszsegugyi, Kereskedelmi es Szolgaltato Kft., Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz, Szombathely
- India (11):
  - Mavani Research Center, Ahmedabad, Gujarat
  - Shalby Hospital, Ahmedabad, Gujarat
  - Government Medical College Thiruvananthapuram, Thiruvananthapuram, Kerala
  - Noble Hospital, Hadapsar, Maharashtra
  - P. D. Hinduja Hospital and Medical Research Centre, Mumbai, Maharashtra
  - Shree Siddhivinayak Maternity & Nursing Home, Nashik, Maharashtra
  - Max Super Speciality Hospital, Saket, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - Madras Medical College, Chennai, Tamil Nadu
  - Institute of Post-Graduate Medical Education and Research, Kolkata, West Bengal
  - Osmania General Hospital, Telangana
- Israel (12):
  - Assuta Ashdod Public Hospital (R.A), Ashdod
  - Barzilai Medical Center | Department of Nephrology and Hypertension, Ashkelon
  - Clalit Health | Soroka Medical Center - Internal Medicine Department, Beersheba
  - Rambam Health Corporation, Haifa
  - Meir Medical Center, Kfar Saba
  - Health Corporation of Galilee Medical Center, Nahariya
  - Rabin Medical Center | Beilinson Hospital - Internal Medicine C Department, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Poria Medical Center | Nephrology and Hypertension Department, Tiberias
  - Shamir Medical Center (Assaf Harofeh), Ẕerifin
- Italy (12):
  - A.O.U. Universita' Degli Studi Della Campania Luigi Vanvitelli - Nefrologia, Napoli, Campania
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS_Policlinico Sant'Orsola - Nefrologia, Dialisi e Trapianto, Bologna, Emilia-Romagna
  - Azienda Ospedaliero Universitaria di Modena_Policlinico - Nefrologia, Dialisi e Trapianto di Rene, Modena, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Parma - SC Nefrologia, Parma, Emilia-Romagna
  - Azienda USL IRCCS di Reggio Emilia_Arcispedale Santa Maria Nuova - S.C. Nefrologia e Dialisi, Reggio Emilia, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Nefrologia, Rome, Lazio
  - Azienda Socio Sanitaria Territoriale Della Brianza_Ospedale Pio XI - Nefrologia e Dialisi, Desio, Lombardy
  - Azienda Socio Sanitaria Territoriale Ovest Milanese_Legnano - Nefrologia e Dialisi, Legnano, Lombardy
  - Istituti Clinici Scientifici Maugeri S.p.A._Pavia - Nefrologia, Pavia, Lombardy
  - Istituto Ricerche Farmacologiche Mario Negri - Unità Operativa Complessa Malattie Renali, Ranica, Lombardy
  - Azienda Socio Sanitaria Territoriale Rhodense, Rho, Lombardy
  - Azienda Ospedaliera Per L'Emergenza Cannizzaro - Nefrologia e Dialisi, Catania, Sicily
- Japan (41):
  - Chubu Rosai Hospital, Nagoya, Aichi-ken
  - Daido Clinic, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Kainan Hospital, Yatomi, Aichi-ken
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Aso Iizuka Hospital, Iizuka, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - JCHO Kyushu Hospital, Kitakyushu, Fukuoka
  - Central Japan International Medical Center, Minokamo, Gifu
  - Kobe University Hospital, Kobe, Hyōgo
  - Hyogo Prefectural Nishinomiya Hospital, Nishinomiya, Hyōgo
  - JA Toride Medical Center, Toride, Ibaraki
  - Tsuchiura Kyodo General Hospital, Tsuchiura, Ibaraki
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - National Hospital Organization Kanazawa Medical Center | Clinical Trial Management Office, Kanazawa, Ishikawa-ken
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Hiratsuka Kyosai Hospital, Hiratsuka, Kanagawa
  - Tokai University Hospital, Isehara, Kanagawa
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Saiseikai Yokohamashi Nanbu Hospital, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Yokohama Sakae Kyosai Hospital, Yokohama, Kanagawa
  - Matsumoto City Hospital, Matsumoto, Nagano
  - Shinshu University Hospital, Matsumoto, Nagano
  - Kawasaki Medical School Hospital, Kurashiki, Okayama-ken
  - Osaka Rosai Hospital, Sakai, Osaka
  - Saitama Medical University Hospital, Irima-gun, Saitama
  - Koshigaya Municipal Hospital, Koshigaya, Saitama
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Tama Medical Center, Fuchū, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - Social Medical Corporation the Chiyukai foundation Fukuoka Wajiro Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Nara Prefecture General Medical Center, Nara
  - Saga-Ken Medical Centre Koseikan, Saga
  - Japanese Red Cross Saitama Hospital, Saitama
- Malaysia (11):
  - Hospital Selayang, Shah Alam, Selangor
  - Hospital Sultan Abdul Halim, Kedah
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Universiti Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuala Pahang
  - Hospital Kajang, Kuala Selangor
  - Hospital Pakar Sultanah Fatimah, Muar town
  - Hospital Tuanku Jaafar | Nephrology Department, Negeri Sembilan
  - Hospital Raja Permaisuri Bainun, Perak
  - Hospital Seri Manjung, Perak
  - Hospital Pulau Pinang, Pulau Pinang
- Mexico (4):
  - Fundacion Cardiovascular de Aguascalientes | Aguascalientes, Mexico, Missing, Aguascalientes
  - SINACOR | Culiacan, Mexico, Culiacán, Sinaloa
  - Sociedad de Metabolismo y Corazon S.C. | Veracruz, Mexico, Puerto de Veracruz, Veracruz
  - Sitio Alfredo Chew Wong | Aguascalientes, Mexico, Aguascalientes
- Portugal (5):
  - Unidade Local De Saúde De Lisboa Ocidental E.P.E., Carnaxide, Lisbon District
  - Centro Hospitalar do Medio Tejo | Unidade de Torres Novas - Nephrology Department, Torres Novas, Santarém District
  - Unidade Local de Saude Almada-Seixal | Hospital Garcia de Orta - Research Department, Almada, Setúbal District
  - Centro Hospitalar de Leiria | Santo Andre Hospital - Research Center, Leiria
  - Centro Hospitalar Universitario de Lisboa Central | Hospital Curry Cabral - Nephrology Department, Lisbon
- Russia (12):
  - First City Clinical Hospital n.a. E.E. Volosevich, Arkhangelsk
  - Izhevsk City Clinical Hospital #9, Izhevsk
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - City clinical hospital n.a. V.V. Vinogradov, Moscow
  - City Hospital #52, Moscow
  - City Clinical Hospital of Emergency Care #1, Omsk
  - Rostov State Medical University, Rostov-on-Don
  - Limited liability company "MK-Med", Saint Petersburg
  - Saratov City Clinical Hospital #9, Saratov
  - City clinical hospital #40 Sestroretsk, Sestroretsk
  - Voronezh Regional Clinical Consultancy-Diagnostic Center, Voronezh
  - Regional Clinical Hospital Yaroslavl, Yaroslavl
- Singapore (5):
  - National University Hospital Medical Centre, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - SingHealth Polyclinics - Pasir Ris, Singapore
  - Khoo Teck Puat Hospital, Singapore
- South Korea (17):
  - Yonsei University Wonju Christian Hospital, Wŏnju, Gang''weondo
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggido
  - Dongguk University Ilsan Hospital, Goyang-si, Gyeonggido
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggido
  - CHA Bundang Medical Center | Nephrology, Seongnam-si, Gyeonggido
  - The Catholic University of Korea, Incheon St.Mary's Hospital, Incheon, Incheon Gwang''yeogsi
  - Kangdong Sacred Heart Hospital, Teugbyeolsi, Seoul
  - The Catholic Univ. of Korea Eunpyeong St. Mary's Hospital, Seoul, Seoul Teugbyeolsi
  - Severance Hospital, Yonsei University Health System - Cardiology, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Inje University Busan Paik Hospital, Busan
  - Chung Nam National University Hospital, Daejeon
  - Ansan Hospital | Nephrology, Gyeonggi-do
  - Samsung Medical Center - Cardiology, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Kangnam Sacred Heart Hospital, Seoul
- Spain (11):
  - Area Sanitaria De Ferrol | Medicina Interna, Ferrol, A Coruña
  - Bellvitge Hospital Universitari | Nefrologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Publico Da Marina | Nefrologia, Burela de Cabo, Lugo
  - Hospital Universitario Central De Asturias | Nefrologia, Alcalá de Henares, Madrid
  - Hospital del Mar | Nephrology Department, Barcelona
  - Hospital Universitari Vall D Hebron | Nefrologia, Barcelona
  - Hospital Universitario Ramon Y Cajal | Medicina Interna, Madrid
  - Hospital Universitario 12 De Octubre | Nefrologia, Madrid
  - Hospital Clinico Universitario De Valencia | Nefrologia, Valencia
  - Hospital Universitario Dr Peset Aleixandre | Nefrologia, Valencia
  - Hospital Universitario Y Politecnico La Fe | Nefrologia, Valencia
- Taiwan (9):
  - National Taiwan University Hospital, Hsin-Chu Branch, Taoyuan District, Hsinchu
  - Far Eastern Memorial Hospital | Nephrology Department, New Taipei City, Taipei
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University | Clinical Research Center, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District
- United Kingdom (6):
  - Barts Health NHS Trust - Royal London Hospital - Nephrology, London, Greater London
  - King's College Hospital NHS Foundation Trust | King's College Hospital - Nephrology Department, London, Greater London
  - Kent and Canterbury Hospital | Renal Research Delivery Team, Canterbury, Kent
  - Sheffield Teaching Hospitals NHS Foundation Trust | Northern General Hospital - NIHR Sheffield Clinical Research Facility, Sheffield, South Yorkshire
  - Cardiff and Vale University Health Board | University Hospital of Wales - Nephrology and Transplant, Cardiff, Wales
  - Gloucestershire Hospitals NHS Foundation Trust | Gloucestershire Royal Hospital - Nephrology, Gloucester

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Ostrominski JW, Filippatos G, Claggett BL, Miao ZM, Desai AS, Jhund PS, Henderson A, Rohwedder K, Brinker MD, Scalise A, Schloemer P, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Rossing P, Ruilope LM, Anker SD, Pitt B, Agarwal R, McMurray JJV, Solomon SD, Vaduganathan M. Effect of Finerenone on Morbidity and Mortality in CKD. J Am Soc Nephrol. 2025 Sep 12. doi: 10.1681/ASN.0000000823. Online ahead of print. No abstract available. PMID 40938666
- [Derived] Zachariah T, Radhakrishnan J. Potential Role of Mineralocorticoid Receptor Antagonists in Nondiabetic Chronic Kidney Disease and Glomerular Disease. Clin J Am Soc Nephrol. 2024 Nov 1;19(11):1499-1512. doi: 10.2215/CJN.0000000000000540. Epub 2024 Jul 22. PMID 39037799